CLINICAL TRIAL: NCT02787317
Title: Bivalirudin in Stable Ischemic Heart Disease Patients Undergoing PCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Chinese PLA General Hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChinaPLA general hospital
Record Dates: First submitted 2016-05-24; First posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Coronary Disease
Keywords: bivalirudin; myocardial injure
MeSH Terms: conditions — Coronary Disease | interventions — bivalirudin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- heparin (Active Comparator): For the heparin group, a bolus dose of 100 U/kg was administered according to current guidelines.
  Interventions: Drug: Heparin
- not prolong infusion Bivalirudin (Experimental): Bivalirudin was given as a bolus of 0.75mg/kg followed by infusion of 1.75mg/kg/h during the PCI procedure .
  Interventions: Drug: bivalirudin
- prolong infusion bivalirudin (Experimental): Bivalirudin was given as a bolus of 0.75mg/kg followed by infusion of 1.75mg/kg/h during the PCI procedure and prolong for 4 hours after procedure.
  Interventions: Drug: bivalirudin

INTERVENTIONS:
Drug: bivalirudin — Bivalirudin is an alternative to heparin in patients undergoing percutaneous coronary intervention.
  Arms: not prolong infusion Bivalirudin; prolong infusion bivalirudin
Drug: Heparin — Heparin is used in patients undergoing percutaneous coronary intervention.
  Arms: heparin

SUMMARY:
Prolonging infusions may decrease myocardial damage associated with bivalirudin use during primary PCI. The investigators hypothesized that continuing the bivalirudin infusion commenced during the procedure at the PCI recommended dose for 4 hours would prevent myocardial damage.

DETAILED DESCRIPTION:
Bivalirudin is widely used as an anticoagulant during percutaneous coronary intervention (PCI) for coronary heart disease. Prolonging infusions may decrease myocardial damage associated with bivalirudin use during primary PCI . However, whether prolonging infusions of bivalirudin could prevent ischemic complications is unknown. The investigators examined the effects of prolonged drug infusion after elective PCI. The investigators hypothesized that continuing the bivalirudin infusion commenced during the procedure at the PCI recommended dose for 4 hours would prevent myocardial damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80 years with stable ischemic heart disease in whom PCI was required.

Exclusion Criteria:

* cardiogenic shock;
* thrombolytic therapy administered before randomization or any anticoagulant administered within 48 hours of randomization;
* active or recent major bleeding or bleeding predisposition;
* major surgery within 1 month;
* clinical syndrome suspicious for aortic dissection, pericarditis, or endocarditis;
* blood pressure higher than 180/110 mm Hg;
* known hemoglobin less than 10 g/dL, platelet count less than 100 × 109/L, aminotransferase level greater than 3 × the upper limit of normal, or creatinine clearance less than 30 mL/min;
* history of heparin-induced thrombocytopenia;
* allergy to any of the study drugs or devices;
* pregnancy or lactation;
* any condition making PCI unsuitable or that might interfere with study adherence; and
* patient unwilling or unable to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1770 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
creatine kinase-MB increase | up to postprocedural 72 hours
  creatine kinase-MB increase >3 times upper limit of normal

SECONDARY OUTCOMES:
bleeding（BARC class） | 30 days and 1 year
  including BARC class 2-5
major adverse cardiac or cerebral events | 30 days and 1 year
  a composite of all cause death, reinfarction, target vessel revascularization or stroke
Net Adverse Clinical Events | 30 days and 1 year
  a composite of all cause death, any myocardial infarction, any target vessel revascularization, stroke or any bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- ChinaPLAGH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Han Y, Guo J, Zheng Y, Zang H, Su X, Wang Y, Chen S, Jiang T, Yang P, Chen J, Jiang D, Jing Q, Liang Z, Liu H, Zhao X, Li J, Li Y, Xu B, Stone GW; BRIGHT Investigators. Bivalirudin vs heparin with or without tirofiban during primary percutaneous coronary intervention in acute myocardial infarction: the BRIGHT randomized clinical trial. JAMA. 2015 Apr 7;313(13):1336-46. doi: 10.1001/jama.2015.2323. PMID 25775052
- [Result] Cortese B, Picchi A, Micheli A, Ebert AG, Parri F, Severi S, Limbruno U. Comparison of prolonged bivalirudin infusion versus intraprocedural in preventing myocardial damage after percutaneous coronary intervention in patients with angina pectoris. Am J Cardiol. 2009 Oct 15;104(8):1063-8. doi: 10.1016/j.amjcard.2009.06.005. PMID 19801025